CLINICAL TRIAL: NCT01050634
Title: Sequencing Of Endocrine Therapy In Post-Menopausal Women With Early Breast Cancer (FAST) a Non-interventional Trial With Aromasin®
Brief Title: Sequencing Of Endocrine Therapy In Post-Menopausal Women With Early Breast Cancer (FAST)
Acronym: FAST
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Other Study IDs: A5991079
Record Dates: First submitted 2010-01-13; First posted 2010-01-15 (Estimated); Results first posted 2010-07-23 (Estimated); Last update posted 2010-07-23 (Estimated); Status verified 2010-06

CONDITIONS: Post Menopausal Women With Early Breast Cancer
Keywords: Aromatase inhibitor; Switch after Tamoxifen; Quality of Life; Safety
MeSH Terms: interventions — exemestane

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observational
  Interventions: Drug: Aromasin (exemestane)

INTERVENTIONS:
Drug: Aromasin (exemestane) — 25mg oral tablet, daily, for >1yr
  Other Names: Aromasin, exemestane

SUMMARY:
Quality of life under therapy with Aromasin® (exemestane) according to IBCSG (International Breast Cancer Study Group) questionnaire.

Change of the endometrium after switching from tamoxifen to Aromasin® (exemestane).

Deeper knowledge of Adverse Events during routine administration.

ELIGIBILITY:
Inclusion Criteria:

* Early Breast Cancer, post-menopausal, 2-3 yrs adjuvant tamoxifen therapy.

Exclusion Criteria:

* Not applicable.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Early Breast Cancer, post-menopausal, 2-3 yrs adjuvant tamoxifen therapy
Sampling Method: Non-Probability Sample
Enrollment: 980 (Actual)
Dates: Start 2005-11; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5991079&StudyName=Sequencing%20Of%20Endocrine%20Therapy%20In%20Post-Menopausal%20Women%20With%20Early%20Breast%20Cancer%20%28FAST%29

RESULTS

PARTICIPANT FLOW:
Groups:
- Aromasin (Exemestane): The recommended dosage of exemestane was 25mg once a day.
Period: Overall Study
Arm/Group | Aromasin (Exemestane)
Started | 980
Received Treatment | 924
Completed | 852
Not Completed | 128
Not completed — Enrolled, but Not Treated | 56
Not completed — Death | 2
Not completed — Adverse Event | 42
Not completed — Lost to Follow-up | 2
Not completed — Other | 21
Not completed — Ongoing at Date of Cut-Off | 5

BASELINE CHARACTERISTICS:
Groups:
- Aromasin (Exemestane): The recommended dosage of exemestane was 25 mg once a day.
Arm/Group | Aromasin (Exemestane)
Number analyzed (Participants) | 924
Age, Customized [Number; unit: Participants]
  18-44 years | 24
  45-64 years | 450
  >= 65 years | 417
  Unspecified | 33
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 924
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in International Breast Cancer Study Group (IBCSG) Linear Analogues Self-Assessment (LASA) Quality of Life (QoL) Core Questionnaire Scores
Description: 10 single-item in LASA format(100mm scale): Physical wellbeing (good to lousy); Mood (happy to miserable); Tiredness, Hot flushes, Feeling sick, Use of arm restricted - all none to a lot; Appetite (good to none); Effort to cope with illness (no effort to great deal of effort); Supported by people (much to not at all); Rating life in current condition (perfect to worst health). Individual items scored by measuring distance in mm between left scale anchor and patient's mark, where best QoL=0mm, worst QoL =100mm, and negative changes from baseline=improvement in QoL.Score range=0-100
Time Frame: Baseline, Month 12
Population: Full Analysis Set (FAS)=Subjects who received at least 1 dose of study treatment and had at least 1 post-baseline efficacy measurement=Number of participants analyzed. Missing values were imputed by last observation carried forward (LOCF). Subjects analyzed for single item (n)=Subjects with Baseline and Final Visit (LOCF) scores for the item
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Aromasin (Exemestane)
Number analyzed (Participants) | 860
mm
  Physical Well-Being (n=773) | -5.82 (23.58)
  Mood (n=775) | -8.37 (21.88)
  Tiredness (n=774) | -8.22 (23.20)
  Appetite (n=776) | -7.04 (21.35)
  Hot Flushes (n=772) | -5.98 (24.65)
  Feeling Sick (Nausea/Vomiting) (n=774) | -2.06 (15.52)
  Effort to Cope with Illness (n=773) | -11.0 (22.95)
  Feel Supported by People Close to You (n=774) | -2.09 (18.23)
  Operation Restricts Use of Arm (n=771) | -4.96 (18.64)
  Imagine Rest of Life in Current Condition (n=767) | -5.42 (17.69)

2. Primary Outcome: Change From Baseline in Thickness of Endometrium
Description: Ultrasound measurement. New derived variable for normalization of endometrium thickness:
  1 = Endometrium thickness <=5mm 0 = Endometrium thickness >5mm
Time Frame: Baseline, Month 12
Population: FAS. Missing values were imputed by LOCF. Number of participants analyzed=Number of subjects with Baseline and Final Visit (LOCF) values.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Aromasin (Exemestane)
Number analyzed (Participants) | 437
mm | -1.1 (6.1)

3. Primary Outcome: Change From Baseline in IBCSG LASA Items Scores - QoL Module 24-26
Description: Assessment of severity of 13 items (Being irritable, Sweats, Vaginal discharge, dryness, and itching/irritation, Sleep disturbance, Feeling dizzy, Headaches, Bone or joint pain, Troubled by weight gain, Loss of sexual interest, Difficulties in becoming aroused - all from none to severe, and Bothered by treatment related difficulties (not at all to severely). Individual items scored by measuring distance in mm between left scale anchor and patient's mark, where no severity=0mm, maximum severity=100mm and negative changes from baseline=lessening of severity.Score range=0-100
Time Frame: Baseline, Month 12
Population: FAS=Number of participants analyzed. Missing values were imputed by LOCF. Number of subjects analyzed for single LASA item (n)=Number of subjects with Baseline and Final Visit (LOCF) scores for the single item.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Aromasin (Exemestane)
Number analyzed (Participants) | 860
mm
  Being Irritable (n=771) | -5.22 (20.58)
  Sweats (Including Night Sweats) (n=771) | -7.44 (23.63)
  Vaginal Discharge (n=766) | -3.45 (17.67)
  Vaginal Dryness (n=765) | -4.98 (26.44)
  Vaginal Itching/Vaginal Irritation (n=765) | -1.70 (20.89)
  Sleep Disturbance (n=769) | -5.35 (22.48)
  Feeling Dizzy (n=768) | -2.42 (19.28)
  Headaches (n=771) | -2.11 (18.97)
  Bone or Joint Pain (n=772) | 1.67 (26.49)
  Troubled by Weight Gain (n=770) | -5.39 (21.69)
  Loss of Sexual Interest (n=741) | -3.25 (25.64)
  Overall Bothered by Treatment (n=718) | -6.59 (22.48)
  Had Difficulties Becoming Aroused? (n=345) | -3.37 (19.94)

4. Primary Outcome: Change From Baseline in 12-Item Short Form Health Survey (SF-12) Summary Subscales (Physical Summary Scale Derived From Items 1-5, 8 and Mental Summary Scale Derived From Items 6, 7, 9-11) Scores
Description: Items: 1.General health 1=poor to 5=excellent 2.Limited moderate activities & 3.Climbing of stairs 1=lot to 3=not at all 4.Accomplished less & 5.Limited in kind of work due to physical health, 6.Accomplished less & 7.Work done less carefully due to emotional problems 1=yes, 2=no 8.Pain interfered with work 1=extremely to 5=not at all 9.Felt calm & 10.Had lot of energy 1=none to 6=all time 11.Felt downhearted & 12.Physical health/emotional problems interfered with social activities 1=all time to 6=none of the time. Higher scores=better QoL, positive changes from baseline=improvement in QoL.
Time Frame: Baseline, Month 12
Population: FAS. Missing values were imputed by LOCF. Number of participants analyzed=Number of subjects with Baseline and Final Visit (LOCF) Scores.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Aromasin (Exemestane)
Number analyzed (Participants) | 758
Scores on a scale
  Mental Summary Scale | 2.93 (8.90)
  Physical Summary Scale | 2.02 (7.14)

5. Primary Outcome: Change From Baseline in IBCSG Vaginal Symptoms - QoL Module 24-26
Description: The 3 LASA items concerning vaginal symptoms (discharge, dryness, itching/irritation) were combined as the sum of these 3 items. Lower scores corresponded to better QoL, with negative changes from baseline corresponding to improvements in vaginal symptoms. Total overall score range=0-300, Best score=0, Worst score=300
Time Frame: Baseline, Month 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Scores on a scale (mm)
Arm/Group | Aromasin (Exemestane)
Number analyzed (Participants) | 756
Scores on a scale (mm) | -10.2 (47.31)

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Observational
Serious Adverse Events (participants affected / at risk) | 11/924
Other Adverse Events (participants affected / at risk) | 82/924
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Observational (N=924)
Cardiac failure (Cardiac disorders) | 1
Gastric ulcer (Gastrointestinal disorders) | 1
Fall (Injury, poisoning and procedural complications) | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 2
Blood pressure increased (Investigations) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Tumour invasion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Carpal tunnel syndrome (Nervous system disorders) | 1
Confusional state (Psychiatric disorders) | 1
Thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Observational (N=924)
Presbyacusis (Ear and labyrinth disorders) | 1
Autoimmune thyroiditis (Endocrine disorders) | 1
Cataract (Eye disorders) | 1
Visual acuity reduced (Eye disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 3
Gastritis (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 1
General physical health deterioration (General disorders) | 1
Oedema (General disorders) | 1
Oedema peripheral (General disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Seasonal allergy (Immune system disorders) | 1
Cystitis (Infections and infestations) | 1
Erysipelas (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Arthropod bite (Injury, poisoning and procedural complications) | 1
Rib fracture (Injury, poisoning and procedural complications) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 21
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 1
Arthropathy (Musculoskeletal and connective tissue disorders) | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 10
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Nodal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Osteopenia (Musculoskeletal and connective tissue disorders) | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 2
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Carpal tunnel syndrome (Nervous system disorders) | 3
Dizziness (Nervous system disorders) | 2
Headache (Nervous system disorders) | 3
Hypoaesthesia (Nervous system disorders) | 1
Memory impairment (Nervous system disorders) | 1
Sensory disturbance (Nervous system disorders) | 1
Visual field defect (Nervous system disorders) | 1
Confusional state (Psychiatric disorders) | 1
Initial insomnia (Psychiatric disorders) | 1
Sleep disorder (Psychiatric disorders) | 1
Thinking abnormal (Psychiatric disorders) | 1
Menometrorrhagia (Reproductive system and breast disorders) | 1
Menopausal symptoms (Reproductive system and breast disorders) | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1
Vulvovaginal dryness (Reproductive system and breast disorders) | 1
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1
Acne (Skin and subcutaneous tissue disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 5
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 2
Menopause (Social circumstances) | 2
Hot flush (Vascular disorders) | 6
Peripheral vascular disorder (Vascular disorders) | 1
Varicose vein (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.